CLINICAL TRIAL: NCT04267094
Title: A Single-center, Multi-scanner, Observational Study to Investigate the Impact of Reduced Radiation Dose and Iterative Reconstruction Algorithms on Coronary Calcium Score in Comparison to the Standard Normal Radiation Dose -Filtered Back Projection Method
Brief Title: Reduced Radiation Dose and IR-impact on Coronary Calcium Quantification
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Science has changed
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Harold Litt, MD, PhD, Associate Professor of Radiology, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 824735
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerotic Plaque
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Iterative reconstruction at reduced radiation dose — Evaluating Agatston coronary calcium score using reduced dose acquisitions reconstructed using iterative reconstruction

SUMMARY:
Evaluation of reduced radiation dose iterative reconstruction reconstructions for calcium scoring compared to full dose filtered back projection reconstructions

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine calcium scoring CT at facilities at the University of Pennsylvania

Exclusion Criteria:

* Patients found to have no coronary calcium on full dose FBP reconstructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Calcium score | immediate
  Calcium score compared to FBP full dose recon

SECONDARY OUTCOMES:
Risk stratification | immediate
  Cardiovascular risk stratification group of reduced dose IR vs. full dose FBP

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States